CLINICAL TRIAL: NCT02623686
Title: What is the Effect of an Aromatherapy Intervention on Sleep in the ICU? An Exploratory Study
Brief Title: The Effect of an Aromatherapy Intervention on Sleep in the ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCR 4308
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Sleep Deprivation
Keywords: Sleep; ICU; Massage Therapy; Inhalation Patch
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aroma group (Experimental): * two massages delivered within a two day period
  * the patient will choose the essential oils used from blend A and blend B (if no choice is made, therapist will choose blend A and B alternately). One drop of the essential oil blend will be added to 5 mls of grapeseed base oil.
  * an Inhalation Patch with the same blend of oils as used in the massage will be left by the therapist for use on each of the two nights following the aromatherapy massage intervention. Its use will be explained to the patient and to the member of nursing staff. The Inhalation Patch will be applied to the patient's upper chest when it is time to sleep at approximately 11 pm and will be removed the following morning at approximately 6 am.
  Interventions: Other: Aroma Therapy Massage and Inhalation Patch
- Control Group (No Intervention): Normal Care

INTERVENTIONS:
Other: Aroma Therapy Massage and Inhalation Patch
  Arms: Aroma group

SUMMARY:
It is known from the literature that patients in the Intensive Care Unit do not get enough sleep impacting on short and longterm recovery (Tembo & Parker, 2009; Bihari et al, 2012; Kamdar et al, 2012). The use of non-pharmacological interventions such as massage with essential oils is supported by the literature as being useful in encouraging sleep (Richards et al, 2003; Matthews, 2011). Over 30% of cancer patients are accessing complementary therapies such as these (Rees et al, 2000; Lewith et al, 2002). We propose investigating whether aromatherapy massage and the use of essential oils in the form of an Inhalation Patch (Bioesse TM) prove to be a useful intervention for improving patient sleep whilst on the critical care unit.

DETAILED DESCRIPTION:
A search of the literature shows that patients in the ICU specifically do not get enough sleep. The causes for this are multifactorial and include nursing and medical procedures, pain, discomfort, anxiety, stress, mechanical ventilation, the ICU environment including noise and light, pharmacological agents and severity of underlying disease (Tembo & Parker, 2009; Bihari et al, 2012; Kamdar et al, 2012). Sleep disruption, along with inability to communicate and limitations on visiting, were rated as stressors by ICU patients (Nelson et al, 2001). The effects of poor sleep are deleterious, impacting on patients' recovery both within the ICU (Tembo & Parker, 2009; Bihari et al, 2012) and subsequently after discharge (Kamdar et al 2012). Measurements on mechanically ventilated patients receiving continuous intravenous sedation showed disturbed Circadian timing, lack of REM sleep and absent EEG features of the alternation of wake and sleep states, suggesting that these patients may be continuously sleep deprived which could exacerbate their condition and compromise their recovery (Gehlbach et al, 2012). There is a preponderance of evidence suggesting that sedation practices may impact a range of adverse outcomes; novel strategies to combat patient symptomatology through non-pharmacologic means are to be encouraged (Millelsen & Schweickert, 2013).Furthermore, the positive effect on anxiety of therapeutic touch using massage on ICU patients has been demonstrated previously in two RCTs (Henricson et al, 2008; Lindgren et al, 2013).The use of non-pharmacological strategies to encourage sleep is suggested by a number of authors (Gosselink et al, 008; Matthews, 2011; Kamdar et al, 2012). Richards (1998) found back massage useful for promoting sleep in critically ill older men; Nerbass et al (2010) found massage improved sleep post coronary artery bypass graft surgery;Soden et al (2004) found sleep scores of palliative care patients with cancer significantly improved with aromatherapy massage and massage alone, despite the fact that the massage interventions were given in the morning. Sleepdisruption can be exacerbated by factors such as pain, anxiety and stress (Kamdar et al, 2012). Massage may influence sleep partly because of its effects on these symptoms; a review by Ernst (2009) concluded that massage may help with symptom control including the reduction of anxiety and pain in cancer palliation and supportive care.Stringer et al (2008) found a single session of massage for isolated hematology patients undergoing intensive chemotherapy brought a significant reduction in cortisol with an accompanying improvement in psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* any NHS patient with cancer admitted to the CCU during the period of the study
* aged 18 years or over
* who wishes to take part in the study

Exclusion Criteria:

* expected length of stay < 4 days
* habitual use of sleep medication more than 3 times per week
* no sleep meds/hypnotics allowed during study period
* no sedation during intervention period (propofol; clonidine; midazolam)
* extensive brain metastases/hypoxic or traumatic brain injury
* sleep apnoea
* excessive alcohol consumption >50 units/week (ascertained via notes)
* extensive wound/skin damage that precludes massage (e.g. drug-related bullae/skin desquamation)
* neuromuscular blockade
* any normal massage contraindications including: severe respiratory or hemodynamic instability, GCS <7*, ICP <20* mmHg, no contraindication for changing in body position (including active significant bleeding etc)
* allergies to the use of essential oils, either on the skin or inhaled, precluding the use of both of the study blends
* allergy to base (grapeseed) oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
• Differences in RCSQ patient scores | 24 months

SECONDARY OUTCOMES:
• Difference in BIS scores | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, London, United Kingdom